CLINICAL TRIAL: NCT07405541
Title: Knowledge of Periodontitis and Its Impact on Periodontal Health: A Comparative Observational Study in Final-Year Dentistry and Psychology Students
Brief Title: Knowledge of Periodontitis and Its Relation to Periodontal Health
Status: Not yet recruiting | Type: Observational
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Sponsor
Other Study IDs: TFG_25-26151.0; TFG_25-26151.0 (Other: Universitat Internacional of Catalunya)
Record Dates: First submitted 2026-01-26; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Presence of Periodontal Disease; Knowledge of Periodontal Disease
Keywords: knowledge; periodontitis; periodontal disease; periodontal diagnosis; dental students
MeSH Terms: conditions — Periodontitis; Periodontal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- students of undergraduate program of dentistry: students of undergraduate program of psychology

SUMMARY:
This study aims to evaluate the level of knowledge regarding periodontal disease and its association with periodontal health status among health sciences students. An observational, cross-sectional, analytical, and comparative design will be conducted involving two cohorts: final-year Dentistry students and Psychology students from the Universitat Internacional de Catalunya (UIC).

A total of approximately 60 participants (30 per group) will be recruited using stratified random sampling. Eligible participants must be at least 18 years old and provide written informed consent. Students who have received periodontal treatment within the previous six months, present uncontrolled systemic diseases, or are pregnant or breastfeeding will be excluded.

Data collection will take place during a single clinical visit between January and April 2026 and will consist of two phases. First, participants will complete a validated Knowledge, Attitudes, and Practices (KAP) questionnaire assessing understanding of periodontitis, attitudes toward oral health, and daily oral hygiene behaviors. Knowledge scores will be categorized into low, medium, and high levels. Second, a comprehensive periodontal examination will be performed by a certified periodontist under standardized conditions, including plaque index, bleeding on probing, probing depth, gingival margin position, clinical attachment loss, and radiographic assessment. Periodontal status will be classified according to the 2018 EFP/AAP classification system using staging and grading criteria.

The primary outcome is the presence of periodontal disease (gingivitis or periodontitis). The main independent variable is the level of knowledge about periodontitis. Covariates include age, sex, oral hygiene habits, smoking status, perceived stress, and self-reported systemic conditions.

Statistical analysis will be conducted using SPSS, Stata, or R software. Descriptive statistics will summarize participant characteristics. Bivariate analyses will assess associations between knowledge level and periodontal disease using chi-square tests and appropriate parametric or non-parametric comparisons. Multivariate binary logistic regression will be applied to evaluate whether lower knowledge levels are independently associated with a higher prevalence of periodontal disease, adjusting for relevant covariates. Statistical significance will be set at p < 0.05.

The study will be conducted following ethical approval from the UIC Research Ethics Committee. Participation will be voluntary, confidentiality will be ensured through anonymized data handling, and participants diagnosed with periodontal disease will be referred for appropriate periodontal care.

DETAILED DESCRIPTION:
Periodontal disease (PD) is defined as a chronic, multifactorial inflammatory disease, characterized by the progressive destruction of the supporting tissues of the teeth. Its development mainly depends on two essential factors: the accumulation of bacterial biofilm and the host's immunoinflammatory response to pathogenic microorganisms. However, other factors also contribute to the onset and progression of the disease, both intraoral and extraoral, including poor oral hygiene, inadequate or harmful dietary habits, and various systemic factors.

The host response to bacterial invasion triggers a series of local inflammatory processes that manifest clinically through signs such as edema, erythema, and gingival bleeding. These manifestations not only affect the oral cavity but may also significantly influence overall systemic health, as PD has been associated with multiple systemic diseases, including diabetes mellitus, cardiovascular diseases, obesity, and pregnancy-related complications. Several studies have shown that the relationship between PD and these conditions is bidirectional: periodontal disease may exacerbate or predispose individuals to these pathologies, while, in turn, these conditions may worsen the progression of PD.

At a global level, PD is recognized as the sixth most prevalent disease worldwide, highlighting the importance of timely and appropriate diagnosis and treatment. In this regard, the American Academy of Periodontology (AAP) and the European Federation of Periodontology (EFP) have proposed an updated classification of periodontal diseases, aimed at enabling more individualized diagnosis and more precise treatment planning. Among the most relevant changes are the redefinition of diagnostic criteria for gingivitis based on objective clinical signs, and the introduction of the concepts of staging and grading, which take into account disease severity, extent, and rate of progression.

Furthermore, this classification acknowledges that certain systemic conditions-such as diabetes mellitus and smoking-modify the grade of the disease, directly influencing treatment planning and the clinical prognosis of each patient.

Regarding therapeutic management, the literature emphasizes that prevention is the most effective measure to reduce the high prevalence of PD. Prevention is based on risk factor control and early detection of initial signs and symptoms. Adequate preventive strategies help avoid frequent complications such as dental sensitivity, halitosis, tooth mobility, and tooth loss, as well as reduce the impact of PD on various systemic diseases.

Healthcare professionals play an essential role in this preventive process, as they are often the first to identify gingival alterations or early signs of inflammation. Therefore, maintaining up-to-date knowledge of periodontal health is fundamental to improving early detection, patient education, and interdisciplinary intervention.

Within this context, the present study proposes the development of an assessment instrument to evaluate knowledge of periodontal health. This instrument focuses on three main aspects:

Identification of the clinical signs of the disease. Recognition of etiological and risk factors. Understanding of the relationship between PD and systemic diseases. The general objective of the study is to determine the level of knowledge regarding periodontal health among health sciences students through the application of a concise, specific, and effective questionnaire to measure their understanding of PD and its interrelationship with systemic health, as well as to evaluate whether the level of knowledge is associated with students' periodontal health status and/or their daily oral hygiene practices, with the aim of implementing educational measures in dentistry across different health sciences degree programs.

2. Background and Current State of the Topic Periodontitis is a chronic inflammatory disease that leads to the loss of dental supporting tissues and may negatively affect general health. Knowledge and oral hygiene practices play a key role in its prevention. Comparing Dentistry students, who receive more extensive training in oral health, with Psychology students allows for the analysis of whether knowledge levels are related to the observed prevalence of periodontal disease, thereby helping to guide interdisciplinary educational interventions.

3. Objectives

Primary objective:

To evaluate the level of knowledge regarding periodontal disease among Dentistry and Psychology students.

To quantify the level of knowledge, attitudes, and practices (KAP) in each group.

Secondary objectives:

To analyze the prevalence of gingivitis and/or periodontal disease in each cohort.

To compare prevalence between both cohorts and estimate the association after adjusting for covariates (age, sex, smoking status, socioeconomic level, medication use, toothbrushing frequency, dental floss use, and relevant systemic diagnoses).

To propose educational recommendations based on the study findings.

Study Design An observational, cross-sectional, analytical, and comparative study will be conducted to evaluate the association between the level of knowledge about periodontitis and the prevalence of periodontal disease in two cohorts: final-year undergraduate students in Dentistry and Psychology at the Universitat Internacional de Catalunya (UIC).

Population and Sample

1. Target population University students enrolled in the Dentistry and Psychology degree programs at the Universitat Internacional de Catalunya during the current academic year.
2. Sampling A randomized and stratified sampling method will be used, considering the two degree programs as strata. A total of 60 participants is expected to be included (30 per group), although this number may be adjusted depending on availability and the population size of each cohort.
3. Inclusion criteria Students enrolled in the Dentistry or Psychology degree programs at UIC. Age ≥ 18 years. Voluntary agreement to participate through signed informed consent.
4. Exclusion criteria Periodontal treatment within the previous 6 months. Presence of uncontrolled systemic diseases that may affect periodontal status (e.g., uncontrolled diabetes mellitus, immunodeficiencies).

   Pregnancy or breastfeeding, if considered relevant according to the Ethics Committee due to potential hormonal alterations affecting periodontal health.

   Withdrawal or refusal of informed consent at any stage of the study. Study Phases and Data Collection

   Data collection will be carried out in two main phases:

   Phase 1: KAP Questionnaire Administration

   A Knowledge, Attitudes, and Practices (KAP) questionnaire, previously adapted and validated in Spanish, will be administered to assess:

   Knowledge regarding periodontitis (etiology, clinical signs, and consequences). Attitudes toward oral health and preventive behaviors. Oral hygiene practices and frequency of dental visits. The questionnaire will be self-administered in digital or paper format, depending on logistical feasibility. It will be completed on the same day as the periodontal examination, in the university dental clinic under the supervision of the principal examiner (PDI) and secondary examiner (IV), in order to minimize potential bias.

   Knowledge-related items will be quantitatively scored and subsequently categorized into three levels: low, medium, and high.

   Phase 2: Clinical Periodontal Examination Each participant will undergo a comprehensive periodontal examination performed by a qualified professional holding the European Board in Periodontology certification (PDI), under standardized biosafety conditions.

   A calibrated millimeter periodontal probe will be used to record the following variables through a full-mouth periodontal chart:

   Plaque Index:

   Assesses the presence or absence of dental plaque on each disclosed tooth surface.

   Plaque Index (%)

   = Number of surfaces with plaque Total number of examined surfaces

   × 100 Plaque Index (%)= Total number of examined surfaces Number of surfaces with plaque
   * 100

   Bleeding on probing:

   Presence or absence of bleeding following probing. 0 = no bleeding 1 = bleeding Bleeding percentage = Number of bleeding sites Total number of examined sites

   × 100 Bleeding percentage= Total number of examined sites Number of bleeding sites

   ×100

   Probing depth (PD):

   Measurement of periodontal pocket depth in millimeters using a calibrated probe.

   Gingival margin position:

   Normal position coinciding with the cemento-enamel junction (CEJ): GM = 0 mm Gingival recession (margin apical to the CEJ): positive value (+) Gingival enlargement (margin coronal to the CEJ): negative value (-)

   Clinical attachment loss (CAL):

   CAL

   = Probing depth

   + Gingival margin position CAL=Probing depth+Gingival margin position Full-mouth radiographic series The assessment will allow classification of participants according to the 2018 periodontal disease classification developed by the European Federation of Periodontology (EFP) and the American Academy of Periodontology (AAP).

   Periodontal Diagnosis Plaque-associated gingival diseases Gingival inflammation caused by bacterial plaque accumulation; reversible with adequate plaque control.

   Non-plaque-induced gingival diseases A heterogeneous group of lesions of genetic, infectious, inflammatory, traumatic, or neoplastic origin.

   Periodontitis

   A diagnosis of periodontitis will be established when:

   Interdental clinical attachment loss is detected in at least two non-adjacent teeth, or Clinical attachment loss of ≥ 3 mm is present at an oral site with probing depth ≥ 3 mm in two or more teeth.

   Periodontitis will be classified using a multidimensional approach based on staging (severity and extent) and grading (risk and rate of progression).

   Stages of Periodontitis

   Staging is based on disease severity and treatment complexity:

   Stage I - Initial periodontitis:

   Radiographic bone loss confined to the coronal third of the root and CAL of 1-2 mm.

   Stage II - Moderate periodontitis:

   Radiographic bone loss in the coronal third and CAL of 3-4 mm.

   Stage III - Severe periodontitis:

   Radiographic bone loss extending to the middle third of the root and CAL ≥ 5 mm, with potential loss of up to four teeth due to periodontal causes.

   Stage IV - Advanced periodontitis:

   Radiographic bone loss extending to the apical third of the root and CAL ≥ 5 mm, with risk of losing five or more teeth and severe masticatory dysfunction.

   Grades of Periodontitis

   Grading reflects the rate of disease progression and future risk, considering modifying factors such as smoking and diabetes mellitus:

   Grade A - Slow progression:

   Favorable response to treatment and minimal risk factors.

   Grade B - Moderate progression:

   Moderate risk and predictable treatment response.

   Grade C - Rapid progression:

   High risk of disease progression and less predictable treatment outcomes, commonly associated with significant risk factors such as heavy smoking.

   Study Timeline

   The study will be conducted in two phases during a single clinical appointment:

   Phase I: Questionnaire administration Phase II: Periodontal examination Data collection will take place between January 2026 and April 2026. Ethical Considerations The study protocol will be submitted for approval to the Research Ethics Committee of the Universitat Internacional de Catalunya.

   All participants will provide written informed consent. Participation will be entirely voluntary, with the right to withdraw at any time without consequences.

   Confidentiality will be ensured through anonymous coding and secure data storage, in accordance with current data protection regulations (Organic Law on Personal Data Protection and Guarantee of Digital Rights - LOPDGDD).

   The study is considered minimal risk, limited to mild discomfort during periodontal probing, with possible bleeding in cases of gingival inflammation.

   Participants presenting signs of periodontal disease will be informed and referred to the Department of Periodontology for appropriate evaluation and treatment.

   6. Results Analysis Study Variables

a) Dependent variable: Level of knowledge about periodontitis (derived from the KAP questionnaire). b) Main independent variable: Presence of periodontal disease (clinically diagnosed gingivitis or periodontitis).

c) Covariates: Age (years, quantitative variable). Sex (male/female/other). Oral hygiene habits (toothbrushing frequency, dental floss use, mouthwash use). Smoking status (smoker/non-smoker, daily consumption). Perceived stress (measured using a subjective scale). Presence of self-reported systemic diseases (diabetes, cardiovascular diseases, etc.).

Statistical Analysis Data will be processed and analyzed using statistical software such as SPSS, Stata, or R.

Descriptive analysis Absolute and relative frequencies will be calculated for categorical variables. Mean, median, and standard deviation will be calculated for quantitative variables.

Bivariate analysis The Chi-square test will be used to explore the association between level of knowledge and the presence of periodontal disease.

Student's t-test or Mann-Whitney U test will be applied to compare mean values between groups, depending on data distribution.

Multivariate analysis A binary logistic regression model will be applied to evaluate whether a low level of knowledge is significantly associated with a higher prevalence of periodontal disease, adjusting for potential confounders (age, sex, smoking status, etc.).

A level of statistical significance of p < 0.05 will be considered.

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled in the Dentistry or Psychology degree programs at UIC.
* Age 18 years or older.
* Voluntary agreement to participate through signed informed consent.

Exclusion Criteria:

* Periodontal treatment within the past 6 months.
* Presence of uncontrolled systemic diseases that may affect periodontal status (e.g., uncontrolled diabetes, immunodeficiencies).
* Pregnancy or breastfeeding, if deemed relevant by the Ethics Committee due to potential hormonal alterations affecting periodontal health.
* Withdrawal or refusal of consent at any stage of the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Undergraduate students from the University Internacional of Catalunya. Dentistry and Psychology, from a random sample
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Periodontal knowledge was assessed using the following questionnaire items: knowledge of periodontitis, about etiology, symptoms, risk factors, self reported symptoms. | March 2026 to June 2026
  An overall periodontal knowledge score was constructed using ten questionnaire items covering awareness of periodontal disease, causes, symptoms, risk factors, and common misconceptions. Each correct response was awarded one point, yielding a total score from 0 to 10. Based on this score, participants were categorized as having low (0-3 points), moderate (4-7 points), or high (8-10 points) levels of periodontal knowledge. This categorization allowed a simplified and interpretable assessment of periodontal knowledge for statistical analysis.

SECONDARY OUTCOMES:
Full periodontal diagnosis | March 2026 to June 2026
  Plaque Index (PI) Plaque accumulation was assessed as a percentage of teeth with plaque. Each tooth was examined at six sites. The presence or absence of plaque was recorded at each site. The plaque index was calculated as the percentage of sites with plaque relative to the total number of examined sites.
  Bleeding Index (Bleeding on Probing, BOP) Bleeding on probing was evaluated at six sites per tooth using a periodontal probe. The bleeding index was expressed as the percentage of bleeding sites in relation to the total number of examined sites.
  Probing Pocket Depth (PPD) Probing pocket depth was measured in millimeters at six sites per tooth using a standardized periodontal probe. Mean probing depth values were calculated per patient.
  Tooth mobility. presence or absence Gingival Recession It was measured in millimeters as the distance from the cementoenamel junction (CEJ) to the gingival margin at the same six sites per tooth. Recession values were recorded in % per patient

IPD SHARING:
Plan to Share IPD: Undecided